CLINICAL TRIAL: NCT01918241
Title: Saftey and Efficacy Phase II Study of Pegfilgrastim in Preventing Chrmotherapy-induced Neutropenia
Brief Title: Saftey and Efficacy of Pegfilgrastim in Preventing Chrmotherapy-induced Neutropenia
Acronym: PEG-rhG-CSF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Jiuyuan Gene Engineering Co. Ltd., (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Jiangsu Cancer Institute & Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Wuhan TongJi Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Shandong Cancer Hospital and Institute (Other); Changsha Central Hospital (Other); Yangzhou No.1 People's Hospital (Other); Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY062013B
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Neutropenia
Keywords: Pegylation; G-CSF; Efficacy; Satety
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- pegfilgrastim,30mcg/kg (Experimental): On the 3rd day and 6th day in Cycle 2, mean after 48h and 120h of chemotherapy, subjects will be received PEG-rhG-CSF(sc) in a fixed time(9:00±30 min), and the dosage is 30 mcg/kg.
  Interventions: Drug: pegfilgrastim,30mcg/kg
- pegfilgrastim, 60mcg/kg (Experimental): On the 3rd day in Cycle 2, mean after 48h of chemotherapy, subjects will be assigned to PEG-rhG-CSF(sc, single) in a fixed time(9:00±30 min), and the dosage is 60 mcg/kg.
  Interventions: Drug: pegfilgrastim, 60mcg/kg
- pegfilgrastim,100mcg/kg (Experimental): On the 3rd day in Cycle 2, mean after 48h of chemotherapy, subjects will be assigned to PEG-rhG-CSF(sc, single) in a fixed time(9:00±30 min), and the dosage is 100 mcg/kg.
  Interventions: Drug: pegfilgrastim, 100mcg/kg
- filgrastim,5mcg/kg (Experimental): On the 3rd day in Cycle 2, mean after 48h of chemotherapy, subjects will be assigned to controlled group with rhG-CSF(sc, once a day) in a fixed time(9:00±30 min), and the dosage is 5mcg/kg, rhG-CSF must be injected for a continous 14 days, or twice observed the results for ANC from the nadir to counts≥5.0×10^9/L, but at least 7 days.
  Interventions: Drug: filgrastim, 5mcg/kg

INTERVENTIONS:
Drug: pegfilgrastim,30mcg/kg — Two doses SC injection of 30 mcg/kg at postchemotherapy 48hr and 120hr in cycle 2.
  Other Names: PEG-rhG-CSF,30mcg/kg
  Arms: pegfilgrastim,30mcg/kg
Drug: pegfilgrastim, 60mcg/kg — Single SC injection of the appropriate dose of drug ranging from 60 mcg/kg to 100 mcg/kg at postchemotherapy 48hr in cycle 2.
  Other Names: PEG-rhG-CSF,60mcg/kg
  Arms: pegfilgrastim, 60mcg/kg
Drug: pegfilgrastim, 100mcg/kg — Single SC injection of the appropriate dose of drug ranging from 60 mcg/kg to 100 mcg/kg at postchemotherapy 48hr in cycle 2.
  Other Names: PEG-rhG-CSF,100mcg/kg
  Arms: pegfilgrastim,100mcg/kg
Drug: filgrastim, 5mcg/kg — At least 7 days SC injection of 5 mcg/kg at postchemotherapy 48hr in cycle 2.
  Other Names: rhG-CSF,5mcg/kg
  Arms: filgrastim,5mcg/kg

SUMMARY:
This study will assess the Efficacy and Safety of different doses of PEG-rhG-CSF and a single-dose of G-CSF in Preventing Chemotherapy-induced Neutropenia.

DETAILED DESCRIPTION:
The study consist of a screening period and a 21-day chemotherapy period of the same chemotherapy treatment cycle(s).Screening the subjects according to the inclusion criteria and exclusion criteria before 2 weeks of chemotherapy, and the screening successfully patients will be eligible for this study. The 1st chemotherapy treatment cycle defined as subjects screening period, subjects will be treated with the TC or EC regimen on the 1st day, aiming to screen out Chemotherapy-induced Neutropenia of ≥grade 3 (ANC<1.0×10^9/L) who can have the eligible to enter the 2nd chemotherapy treatment cycle, otherwise to quit the study. On the 1st day in cycle 2, subjects will be treated with the same regimen as the 1st chemotherapy treatment cycle, and be received the test drugs or controlled from the 3rd day to observe the efficacy and safety.

【Primary Outcome Measures】:

• Duration of ≥grade 3 neutropenia in cycle 2

【Secondary Outcome Measures】:

* Incidence of ≥grade 3 neutropenia induce;
* Incidence of febrile neutropenia;
* Duration for ANC from chemotherapy finished to ANC nadir and the minimum ANC ;
* Duration for ANC recovery from nadir to 2.0×10^9/L.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-70 years；
* Comfirmed advanced tumor patients by histopathological with regarding initialtreatment or adjuvant, or neoadjuvant chemotherapy,suitable for chemotherapy with canboplatin combined with taxol or cyclophosphamide combined with pharmorubicin in the opinion of the investigator；
* Performance status（EOCG）≤1；
* Normal human peripheral blood are eligible for the chemotherapy, WBC≥3,500 per cubic millilit, ANC ≥ 1,500 per cubic milliliter, PLT ≥ 100,000 per cubic milliliter；
* Normal ECG examination；
* Without liver metastasis patients: the level of ALT、TBIL、AST were in the 2.5 times of upper normal limit; Liver metastasis patients: the level of ALT、TBIL、AST were in the 5 times of upper normal limit;
* Renal function indices：the level of Cr、BUN were bothe in the 1.25 times of upper normal limit;
* Life expectancy >3 months;
* Signed informed consent.

Exclusion Criteria:

* Be treated with radiotherapy in nearly 4 weeks(not included local radiotherapy for the bone metastasis);
* Be treated with hemopoietic stem cell transplantation or bone marrow transplant；
* Not adequately controlled infections(e.g. ANC ≥ 12,000 per cubic milliliter,temperature > 38.2℃)
* Evidence of metastatic disease in bone marrow,or with other malignant tumors （not included cured basal cell carcinoma and endometrial carcinoma）；
* Subjects with unconscious or symptomatic brain metastases；
* Subjects with serious heart、liver and renal disease;
* Subjects with serious diabetes or poor control in glycemia;
* Pregnant or breast-feeding period females;
* Be treated with antibiotics in 72 hours or currently being treated with antibiotics;
* Treated with PEG-rhG-CSF in past;
* Participated 3 or more than 3 clinical trials in nearly a year(as subjects) or any clinical trials in nearly 3 months;
* Allergic disorders or allergies subjects or known hypersensitivity to filgrastim or any of the products to be administered during dosing;
* Suspected or comfirmed evidences of drug、treatment of drugs or alcohol abused;
* Serious Neurological disorders that would affect the consent or observation;
* Other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Duration of ≥grade 3 neutropenia in cycle 2 | 21 days

SECONDARY OUTCOMES:
change of Neutropenia and ANC in cycle 2 | 21 days
  1. Incidence of ≥grade 3 neutropenia;
  2. Incidence of febrile neutropenia;
  3. Measurement the duration from chemotherapy finished to the ANC reached the nadir and the value of ANC's nadir;
  4. Time to ANC recovery,the time from chemotherapy administration until the patient's ANC increasd to 2.0*109/L after the expected nadir

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, CAMS, Beijing, China